CLINICAL TRIAL: NCT00877435
Title: Prize Reinforcement Contingency Management for Cocaine Dependence: a 24-week Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Sylvie Petitjean, Dr. phil, University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNF-105314-120675
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Cocaine-related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cognitive behavioral therapy (CBT) + prize-based contingency management (prizeCM)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- 2 (Active Comparator): Cognitive behavioral therapy (CBT)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT)

SUMMARY:
The purpose of this study is to determine whether prize-based contingency management (prizeCM) combined with cognitive behavioral therapy (CBT) is more effective in the treatment of of cocaine-dependent patients compared to CBT only. Patients were randomized to prizeCM + CBT (experimental group) or to CBT (control group) an treated over 24 weeks. It is the first trial of this type in Europe.

ELIGIBILITY:
Inclusion Criteria:

* cocaine dependence, aged 18 or older, other dependences

Exclusion Criteria:

* severe somatic, brain, or psychiatric disease, attention deficit disorders with medication methylphenidate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2013-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
retention in treatment, cocaine abstinence | 24 weeks
  cocaine abstinence: at least 3 consecutive weeks of cocaine abstinence, the maximum number of weeks of continous abstinence and proportions of cocaine-free urine samples during the entire 24-week and at 6-month follow-up.

SECONDARY OUTCOMES:
patients' satisfaction with the therapy, clinical measures | 24 weeks
  patients' satisfaction with prize-based contingency management and with CBT

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie A Petitjean, Dr. phil., Principal Investigator — Psychiatric Hospital of the University of Basel
Locations (2):
- Switzerland (2):
  - Universitäre Psychiatrischen Kliniken, Basel
  - Fondation Phenix, Geneva

REFERENCES:
- See also: Psychiatric Hospital of the University of Basel - Addiction Research Unit — http://www.upkbs.ch